CLINICAL TRIAL: NCT02269527
Title: Effects of an Integrative Music Therapy Program on the Perception of Noise in the SICU: A Patient, Caregiver, and Physician/Nursing Environmental Study
Brief Title: Effects of Live Music on the Perception of Noise in the SICU: A Patient, Caregiver, and Medical Staff Environmental Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Joanne Loewy, Associate Clinical Professor, Icahn School of Medicine at Mount Sinai
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: GCO 16-0936; IRB 088-10 (Other: Beth Israel Medical Center)
Record Dates: First submitted 2014-05-27; First posted 2014-10-21 (Estimated); Last update posted 2024-02-14 (Actual); Status verified 2024-02

CONDITIONS: Pain; Anxiety; Stress
MeSH Terms: conditions — Pain; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Live music (Other): 1-hour live music 5 days/week
  Interventions: Other: Live music

INTERVENTIONS:
Other: Live music — Providing 1-hour live music 5 days/ week.

SUMMARY:
The use of live music in SICU might affect the perception of noise, which may reduce staff's stress level and further decrease the possibility of clinical errors, reduce patient's anxiety and perception of pain as well as increase compliance from patient and family. Live music might also enhance the quality of stay and promote a holistic healing process for the patient.

DETAILED DESCRIPTION:
In this study, the research team is looking at the effect of the live music provided by a trained music therapist, created through incorporating the noises in the SICU - such as the beeping of the machines as part of the elements in the music, to organize the sound environment as well as introducing familiar songs, chosen according to the cultures and ages of the patients, caregivers and staff, to increase a sense of familiarity and comfort. Through the intervention, the research team hope to ameliorate the effects of a noxious sound environment, which may reduce the stress level of the staff and increase their acuity level while decrease patients and caregivers' anxiety level and improve their mood state and the quality of hospitalization

ELIGIBILITY:
Inclusion Criteria:

* SICU patients, caregivers, and physicians/nursing staff

Exclusion Criteria:

* Non-medical Staff

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Actual)
Dates: Start 2010-06; Primary Completion 2020-03-02 (Actual); Study Completion 2020-03-02 (Actual)

PRIMARY OUTCOMES:
Self-report stress level from SICU staff | 6 months
  Environmental music therapy will reduce stress level for SICU staff.
Pre and Post-intervention score on the perception of SICU noises from SICU and Hospital Anxiety and Depression Scale for SICU patients | 1 week
  Environmental Music Therapy will ameliorate the perception of noises and decrease the anxiety level of SICU patients and caregivers
Pre and Post-intervention score on the perception of SICU noises from SICU patients, caregivers | 1 week

CONTACTS AND LOCATIONS:
Overall Officials: Joanne Loewy, DA, Principal Investigator — Mount Sinai Union Square
Locations (1):
- Mount Sinai Beth Israel, New York, New York, United States